CLINICAL TRIAL: NCT04998864
Title: Assessment of Safety and Feasibility of Exablate Blood-Brain Barrier Disruption for the Treatment of High-Grade Glioma in Patients Undergoing Standard Chemotherapy
Brief Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier (BBB) Disruption in GBM Patients
Status: Completed | Type: Observational
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: BT008E
Record Dates: First submitted 2020-07-27; First posted 2021-08-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Glioma, Malignant; Glioblastoma
Keywords: Glioma, MRgFUS, Exablate, TMZ
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Focused Ultrasound (FUS) BBB Disruption: The Exablate Model 4000 Type 2.0 system is intended for use as a tool to induce localized and temporary blood-brain barrier disruption in patients with glioblastoma undergoing standard of care chemotherapy.
  Interventions: Device: Magnetic Resonance guided Focused ultrasound (MRgFUS)

INTERVENTIONS:
Device: Magnetic Resonance guided Focused ultrasound (MRgFUS) — FUS involves the application of acoustic energy at low frequencies from over 1000 individual transducers into distinct body targets.
  Other Names: Exablate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety of the Exablate Model 4000 Type 2.0 used as a tool to disrupt the BBB in patients with high grade glioma undergoing standard of care therapy.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and feasibility of BBB disruption using the Exablate Type 2.0 system in adult patients with glioblastoma (GBM) undergoing adjuvant TMZ chemotherapy, which occurs following maximal safe surgical resection and completion of the initial concurrent radiation-chemotherapy in accordance with the current standard of care

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible for adjuvant TMZ treatment.
2. Men or women age between 18 and 80 years, inclusive.
3. Able and willing to give informed consent.
4. Grade IV glioma (GBM) confirmed Subjects
5. Karnofsky rating 70-100.
6. Able to communicate during the Exablate BBBD procedure.
7. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Evidence of acute intracranial hemorrhage.
2. The subject presents with severe symptoms and signs of increased intracranial pressure
3. Patients with cerebellar or brainstem tumors.
4. Patients with positive HIV status
5. Patients with brain tumors containing 1p/19q chromosomal co-deletion
6. Patient receiving bevacizumab (Avastin) therapy
7. Patients undergoing other concurrent therapies
8. Cardiac disease or unstable hemodynamics
9. Severe hypertension
10. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment
11. History of a bleeding disorder and/or coagulopathy
12. Known sensitivity to gadolinium-based contrast agents
13. Known sensitivity to ultrasound contrast agent
14. Severely impaired renal function
15. Subjects with significant liver dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioblastoma brain tumor who will undergo surgical resection and chemotherapy as standard of care with temozolomide.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Device and procedure related adverse events | Throughout the study, approximately 12 months.
  The number and severity of device and BBB disruption procedure related adverse events will be evaluated and classified according to the CTCAE
Feasibility of repeated BBB disruption will be evaluated through assessment of post-procedure contrast-enhanced magnetic resonance (MR) imaging | At the time of each ExAblate MRgFUS procedure]
  The repeatability of BBB disruption will be evaluated at each of the 6 procedures and will be evaluated through assessment of post-procedure contrast-enhanced MR imaging.

CONTACTS AND LOCATIONS:
Locations (2):
- Fondazione IRCCS Neurologico Carlo Besta, Milan, Italy
- CINAC-Hospital HM Puerta del Sur, Móstoles, Madrid, Spain